CLINICAL TRIAL: NCT06587971
Title: Intensive Treatment on Periodontitis in Aortic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-GSP-QZ-6
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Aortic Valve Stenosis; Periodontitis
MeSH Terms: conditions — Aortic Valve Stenosis; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comprehensive Periodontal Intervention Group (Experimental): Administering the current guideline-recommended comprehensive periodontal treatment protocol to participants, which includes:
  Oral hygiene education: Providing guidance on proper brushing techniques, smoking cessation, dietary control, and blood sugar management.
  Standard periodontal treatment protocol: Administering standard treatments for chronic periodontitis according to the current guidelines, including supragingival scaling, subgingival scaling, root planing, and periodontal flap surgery.
  Interventions: Procedure: Standard periodontal treatment protocol; Behavioral: Oral hygiene education
- Oral hygiene education group (Placebo Comparator): Administering Oral Hygiene Education to Participants. Providing guidance on proper brushing techniques, smoking cessation, dietary control, and blood sugar management.
  Interventions: Behavioral: Oral hygiene education

INTERVENTIONS:
Procedure: Standard periodontal treatment protocol — Administering standard treatments for chronic periodontitis according to the current guidelines, including supragingival scaling, subgingival scaling, root planing, and periodontal flap surgery.
  Arms: Comprehensive Periodontal Intervention Group
Behavioral: Oral hygiene education — Providing guidance on proper brushing techniques, smoking cessation, dietary control, and blood sugar management.

SUMMARY:
The goal of this clinical trial is to determine if standardized periodontal therapy can effectively slow the progression of aortic valve stenosis in adult patients diagnosed with moderate aortic valve stenosis and coexisting gingivitis or mild-to-moderate periodontitis.

The main questions it aims to answer are: Can periodontal therapy slow the progression of aortic valve stenosis? Is chronic periodontitis an independent risk factor for the accelerated progression of aortic valve stenosis? Researchers will compare a group of patients receiving standardized periodontal therapy to a control group receiving only oral hygiene education to see if periodontal treatment results in a slower progression of aortic valve stenosis.

Participants will undergo initial screening to confirm eligibility based on aortic valve peak velocity and periodontal status. They will then be randomly assigned to either the treatment group, which will receive comprehensive periodontal therapy, or the control group, which will receive only oral hygiene education. Participants will be followed up regularly over a 36-month period, with assessments including echocardiograms to monitor the progression of aortic valve stenosis, periodontal examinations to assess oral health status, and blood tests to measure relevant serum biomarkers. The study will also track any cardiovascular events and adverse events related to the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Aortic valve peak velocity (Vmax) between 3.0 and 3.9 m/s.
* Diagnosis of aortic valve stenosis identified as degenerative aortic valve stenosis.
* Presence of gingivitis or mild-to-moderate periodontitis confirmed by periodontal probing or panoramic dental radiography.
* Willingness to participate in the study and signing of informed consent.

Exclusion Criteria:

* End-stage renal disease with eGFR < 15 ml/min/1.73m² (according to the Cockcroft & Gault formula).
* Pregnant, breastfeeding, and women of childbearing age (except those with effective contraception).
* Factors that may affect study follow-up or adherence to periodontal therapy.
* Patients unwilling or unable to undergo comprehensive periodontal treatment.
* Patients who do not consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Composite Major Cardiovascular Events (MACE) Endpoint | From enrollment to the follow-up periods at 12, 24, and 36 months.
  Composite Major Cardiovascular Events (MACE), including:
  1. Hospitalization or emergency/outpatient visits due to heart failure.
  2. Hospitalization or emergency/outpatient visits due to angina.
  3. Hospitalization or emergency/outpatient visits due to syncope.
  4. Cardiovascular death.
  5. Undergoing interventional or surgical valve replacement.
  6. Non-fatal myocardial infarction.
  7. Undergoing percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG).
  8. Ischemic stroke.

SECONDARY OUTCOMES:
Aortic Valve Peak Velocity Change Endpoint | From enrollment to the follow-up periods at 12, 24, and 36 months.
  The difference in the mean change of aortic valve peak velocity before and after the intervention within the control group and the treatment group.
Serum Biomarker Endpoint | From enrollment to the follow-up periods at 12, 24, and 36 months.
  The difference in common serum biomarkers, such as C-reactive protein and interleukin-6, between the control group and the treatment group.
Periodontal Bacterial Biomarker Endpoint | From enrollment to the follow-up periods at 12, 24, and 36 months.
  The difference in the concentration of periodontal bacterial biomarkers between the control group and the treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Erli Zhang, MD, PhD, Study Chair — China National Center for Cardiovascular Diseases; Erli Zhang, MD, PhD, Principal Investigator — China National Center for Cardiovascular Diseases
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No